CLINICAL TRIAL: NCT02894710
Title: Intravenous Lidocaine in Carcinologic ENT Surgery: A Randomized Controlled Trial for Evaluation of Opioid Saving Strategy and Chronic Post-surgical Pain
Brief Title: Intravenous Lidocaine in Carcinologic ENT Surgery: A Trial for Evaluation of Opioid Saving Strategy and Chronic Post-surgical Pain (ELICO)
Acronym: ELICO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL15_0743; 2015-005799-90 (EudraCT Number)
Record Dates: First submitted 2016-08-11; First posted 2016-09-09 (Estimated); Last update posted 2025-10-03 (Actual); Status verified 2025-09

CONDITIONS: Carcinologic Ear, Nose, and Throat (ENT) Surgery
Keywords: postoperative pain; intravenous lidocaine; chronic post-surgical pain; remifentanil; patient controlled analgesia; morphine consumption; ENT surgery
MeSH Terms: conditions — Pain, Postoperative | interventions — Lidocaine; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lidocaine 20mg/ml (Experimental): Patients in Lidocaine group received an intravenous bolus injection of 1,5 mg/kg lidocaine (0,075mL/kg of Lidocaine 20mg/mL) followed by a continuous lidocaine infusion of 2 mg/kg/hr during surgery (0,1mL/kg/hr of Lidocaine 20mg/mL) and 1 mg/kg/hr in recovery room (0,05mL/kg/hr of Lidocaine 20mg/mL).
  Interventions: Drug: Lidocaine 20mg/ml
- Glucose 5% (placebo) (Placebo Comparator): Patients in control group received an intravenous bolus injection of 0,075mL/kg of placebo (Glucose 5%) by a continuous lidocaine infusion of 0,1mL/kg/hr of placebo (Glucose 5%) during surgery and 0,05mL/kg/hr of placebo (Glucose 5%) in recovery room.
  Interventions: Drug: Glucose 5% (placebo)

INTERVENTIONS:
Drug: Lidocaine 20mg/ml — Patients in Lidocaine group received an intravenous bolus injection of 1,5 mg/kg lidocaine (0,075mL/kg of Lidocaine 20mg/mL) followed by a continuous lidocaine infusion of 2 mg/kg/hr during surgery (0,1mL/kg/hr of Lidocaine 20mg/mL) and 1 mg/kg/hr in recovery room (0,05mL/kg/hr of Lidocaine 20mg/mL).
  Arms: Lidocaine 20mg/ml
Drug: Glucose 5% (placebo) — Patients in control group received an intravenous bolus injection of 0,075mL/kg of placebo (Glucose 5%) by a continuous lidocaine infusion of 0,1mL/kg/hr of placebo (Glucose 5%) during surgery and 0,05mL/kg/hr of placebo (Glucose 5%) in recovery room.
  Arms: Glucose 5% (placebo)

SUMMARY:
Lidocaine, local anesthetic used for more than five decades, is being intravenously administered aiming at managing pain in different types of surgeries with promising results. Opioid-induced hyperalgesia need to be considered in ear-nose-throat (ENT) surgery owing to the difficulty of locoregional anesthesia and high level of opioid consumption.

This randomized study aims to compare quality of perioperative analgesia after infusion of intravenous lidocaine during carcinological ENT surgery. The main purpose of this study is to evaluate morphine consumption during the 48 postoperative hours.

Others purposes are evaluation of peroperative remifentanil consumption, morphine consumption during the 24 postoperative hours, chronic post-surgical pain evaluated from 3 to 6 months after carcinologic ENT surgery, and incidence of side effects that can be attributed to lidocaine infusion.

ELIGIBILITY:
Inclusion Criteria:

* Patient undergoing major carcinological ENT surgery (total laryngectomy, oropharyngectomy with or without mandibulotomy, crico-hyoido-epiglotto-pexy, intraoral extended resection, partial laryngectomy, partial pharyngectomy, extended pelvectomy, pelviglossectomy, with or without pectoralis major flap or free flap, with or without lymphadenectomy)
* Patient receiving standardized Patient Controlled Analgesia (PCA)
* Written informed consent

Exclusion Criteria:

* Hypersensitivity to local anesthetics of the amide group,
* Acute porphyria
* Atrioventricular conduction disorders requiring permanent electro-systolic
* Epilepsy not controlled by treatment
* Hepatocellular insufficiency (PT<50%) or cirrhosis
* Systolic heart failure (LVEF <50%)
* Major inflation State
* Hypersensitivity to any component of Glucose 5%
* Treatment with beta-blockers or antiarrhythmic of Vaughan Williams classification
* BMI > 30kg/m2
* Patient already treated for chronic pain with level 3 analgesic or for neuropathic pain
* Pregnant or lactating women
* Refusal to give consent
* Patient under legal protection measure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-12 (Actual)

PRIMARY OUTCOMES:
Total morphine requirement during the first 48 postoperative hours | 48 postoperative hours (H48)
  Standardized patient control analgesia (PCA) devices will be read at the 48th postoperative hour.

SECONDARY OUTCOMES:
Remifentanil peroperative consumption | At the end of surgery (an average of 3 hours et 10 minutes)
  from the beginning of anesthesia to end of surgery
Total morphine requirement | 24 postoperative hours (H24)
  Total morphine requirement during the first 24 postoperative hours.
Evaluation of chronic post-surgical pain | 3 to 6 months after surgery (M3-6)
  Chronic post-surgical pain will be evaluated from 3 to 6 month after surgery by a personal interview of each patient with the french version of McGill pain questionnaire (Questionnaire de Saint-Antoine - version abrégée)
Incidence of side effects that can be attributed to lidocaine infusion | 3 to 6 months after surgery (M3-6)

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Hospices Civils de Lyon / Hôpital de la Croix Rousse, Lyon
  - Centre Léon Bérard, Lyon

REFERENCES:
- [Background] Omar E, Wallon G, Bauer C, Axiotis G, Bouix C, Soubirou JL, Aubrun F. Evaluation of intravenous lidocaine in head and neck cancer surgery: study protocol for a randomized controlled trial. Trials. 2019 Apr 15;20(1):220. doi: 10.1186/s13063-019-3303-x. PMID 30987664
- [Result] Wallon G, Erbacher J, Omar E, Bauer C, Axiotis G, Thevenon S, Soubirou JL, Aubrun F. Effect of intravenous lidocaine on pain after head and neck cancer surgery (ELICO trial): A randomised controlled trial. Eur J Anaesthesiol. 2022 Sep 1;39(9):735-742. doi: 10.1097/EJA.0000000000001712. Epub 2022 Jul 20. PMID 35852564